CLINICAL TRIAL: NCT04887844
Title: Comparison of the Efficacy of Corticosteroid and Local Anesthetic Injections Combined With Conventional Physiotherapy in Patients With Concomitant Pes Anserine Bursitis and Knee Osteoarthritis:
Brief Title: Efficacy of Corticosteroid and Local Anesthetic Injections Patients With Concomitant Pes Anserine Bursitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Mustafa Fatih YAŞAR, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-MFY-01
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Osteoarthritis Knees Both
Keywords: Pain; Knee; Rehabilitation
MeSH Terms: conditions — Pain | interventions — Lidocaine; Adrenal Cortex Hormones; betamethasone dipropionate, betamethasone sodium phosphate drug combination

STUDY DESIGN:
Intervention Model Description: Group I was received physiotherapy+lidocaine injection, Group II was received physiotherapy+betamethasone dipropionate injection, and group III was only received conventional physiotherapy.
Who Masked: Outcomes Assessor
Masking Description: Participant will be evaluated at baseline, 6 weeks later by an another investigator who does not aware of groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): 34 patients who were diagnosed with concomitant knee osteoarthritis and pes anserine bursitis and met inclusion criteria were included in the study. Inclusion criteria were as follows: having stage II-IV knee osteoarthritis along with pes anserine bursitis, duration of symptoms for more than three months, and age between 20 and 70 years. Primary knee osteoarthritis was diagnosed as per American College of Rheumatology (ACR) criteria and graded via Kellgren-Lawrence radiological classification included in this study.
  Interventions: Drug: Lidocaine injection
- Group II (Active Comparator): 34 patients who were diagnosed with concomitant knee osteoarthritis and pes anserine bursitis and met inclusion criteria were included in the study. Inclusion criteria were as follows: having stage II-IV knee osteoarthritis along with pes anserine bursitis, duration of symptoms for more than three months, and age between 20 and 70 years. Primary knee osteoarthritis was diagnosed as per (ACR) criteria and graded via Kellgren-Lawrence radiological classification included in this study.
  Interventions: Drug: Corticosteroid injection
- Group III (Other): 34 patients who were diagnosed with concomitant knee osteoarthritis and pes anserine bursitis and met inclusion criteria were included in the study. Inclusion criteria were as follows: having stage II-IV knee osteoarthritis along with pes anserine bursitis, duration of symptoms for more than three months, and age between 20 and 70 years. Primary knee osteoarthritis was diagnosed as per (ACR) criteria and graded via Kellgren-Lawrence radiological classification included in this study.
  Interventions: Other: Conventional Physical therapy

INTERVENTIONS:
Drug: Lidocaine injection — Lidocaine injection were applied to the most tender point in the pes anserine region by means of the soft tissue infiltration technique only once at the commencement of the treatment period. All injections were performed by the same physician.
  Other Names: Jetokain, Edaka İlaç AŞ, Turkey
  Arms: Group I
Drug: Corticosteroid injection — Corticosteroid injection were applied to the most tender point in the pes anserine region by means of the soft tissue infiltration technique only once at the commencement of the treatment period. All injections were performed by the same physician.
  Other Names: Diprospan, Merck Sharp Dohme Inc., USA
  Arms: Group II
Other: Conventional Physical therapy — The study participants underwent a physiotherapy program that included a one-time 15-minute cold therapy using ice packs and closed-kinetic chain quadriceps strengthening program as follows; isometric quadriceps exercise, isokinetic concentric, and eccentric quadriceps exercises with heel slides and squads. These exercises were repeated ten times a day, seven days per week, for eight weeks in total
  Arms: Group III

SUMMARY:
To evaluate the efficiencies of local corticosteroid injections and local anesthetics in patients with concomitant pes anserine bursitis and osteoarthritis.

DETAILED DESCRIPTION:
Several treatment options have been tried with varying success rates, including nonsteroidal anti-inflammatory drugs, physiotherapy modalities, cold application with ice-packs, and injection of local anesthetics and/or corticosteroids. Despite a relatively high frequency of this painful condition, surprisingly, few studies have evaluated treatment strategies in randomized controlled study design. To the best of our knowledge, no study in the literature made a comparison of the efficacy of local anesthetic and corticosteroid injections in addition to physiotherapy in the treatment of pes anserine bursitis yet. Thus, we aimed to compare the treatment efficacies of physiotherapy alone, physiotherapy + local anesthetic injection, and physiotherapy + local corticosteroid injection in a randomized controlled study design in patients with concomitant osteoarthritis and pes anserine bursitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients having stage II-IV knee osteoarthritis along with pes anserine bursitis
* Symptom onset for more than three months

Exclusion Criteria:

* Patients who underwent knee operations
* had an inflammatory rheumatic disease
* had a history of knee trauma
* had a meniscus tear
* valgus/varus deformity
* received injection treatment to pes anserine bursa during the preceding year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | eight weeks
  We used paper-based VAS to evaluate the baseline severity and changes in the intensity of pain by different interventions in the entire study cohort. The visual analogue scale was devised by Hayes and Patterson and is used to document pain rating. Subjects self-report the intensity of their pain by placing a handwritten mark at one point of the length of a ten-centimeter line. The two ends of the scale line represent "no pain" and "worst pain experienced" at the zero cm and 10th cm of the scale, respectively.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index | eight weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a self-administered questionnaire comprising 24 items in three different domains. The index measure pain, stiffness, and physical functional disability. Pain, stiffness, and physical functional disability subscales comprise five, two, and seventeen questions, respectively. All subscales consist of 5 answer choices, which range from zero, "not present," to four, "very severe."
3-meter walk test | eight weeks
  We used 3MWT to evaluate the walking speed of the study participants. In this test, the individual is instructed to stand up while they are sitting on a chair with arm support. And then, the person is asked to walk as much distance as possible in 3 minutes without running. The walking time is measured in seconds and recorded, and the walking speed is evaluated for the corresponding age group.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Fatih Yaşar, MD, Principal Investigator — Bolu Abant Izzet Baylsa University; Ramazan KURUL, Ph.D, Principal Investigator — Bolu Abant Izzet Baylsa University
Locations (1):
- Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)